CLINICAL TRIAL: NCT02029157
Title: A Phase III Randomized Double-blind, Placebo-controlled Trial of ARQ 197 in Subjects With c-MET Diagnostic-high Inoperable Hepatocellular Carcinoma (HCC) Treated With One Prior Sorafenib Therapy
Brief Title: A Randomized Double-blind, Placebo-controlled Japanese Phase III Trial of ARQ 197 in Hepatocellular Carcinoma (HCC)
Acronym: JET-HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARQ 197-009
Record Dates: First submitted 2013-12-27; First posted 2014-01-07 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — ARQ 197

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARQ 197 (Experimental): Daily oral dose
  Interventions: Drug: ARQ197
- Placebo (Placebo Comparator): Daily oral dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARQ197
  Arms: ARQ 197
Drug: Placebo
  Arms: Placebo

SUMMARY:
The present clinical trial is aiming to evaluate efficacy of ARQ 197 in patients with hepatocellular carcinoma (HCC), who were resistant or intolerable to one systemic chemotherapy regimen including sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form
* ≥20 years old
* Inoperable HCC which is not eligible for locoregional therapy
* Diagnosed as c-Met high in tumor sample
* Radiographic progression is confirmed during or after systemic chemotherapy including sorafenib, or those who are intolerance to the chemotherapy.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) is 0 or 1
* Child-Pugh Class A
* Having measurable target lesions which are defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1,
* Negative pregnancy test results
* Adequate organ function
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* More than 2 prior systemic chemotherapy.
* Prior therapy of c-Met inhibitor (including antibody)
* Any systemic therapy within ≤2 weeks prior to the randomization
* Locoregional therapy within ≤4 weeks prior to randomization.
* Major surgery within ≤4 weeks prior to the randomization
* Concurrent cancer within ≤5 years prior to the randomization
* History of cardiac diseases
* Active clinically serious infections defined as ≥ Grade 3 according to Common Toxicity Criteria for Adverse Effects (CTCAE) 4.0
* Any psychological disorder affecting Informed Consent
* Diagnosis positive for anti-HIV antibody and/or anti-HTLV-1 antibody
* Blood or albumin transfusion within ≤14 days prior to the screening test
* Concurrent interferon therapy against Hepatitis B Virus (HBV)/ Hepatitis C Virus (HCV)
* Symptomatic brain metastases
* History of liver transplantation
* Inability to swallow oral medications
* Confirmed interstitial lung disease
* Pleural effusion and/or clinically significant ascites
* Pregnancy or breast-feeding
* Without consent to effective single or combined contraceptive methods

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2014-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Estimated median of 8-12 weeks in PFS
  Progression-free survival will be compared between ARQ 197 group and Placebo group, to prove the efficacy of ARQ 197 in the population.

SECONDARY OUTCOMES:
Overall survival | Estimated median of 24 weeks in overall survival
  The date of the events was followed every three months after the end of the treatments of the study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Centers in Japan, Tokyo, Japan

REFERENCES:
- [Derived] Kudo M, Morimoto M, Moriguchi M, Izumi N, Takayama T, Yoshiji H, Hino K, Oikawa T, Chiba T, Motomura K, Kato J, Yasuchika K, Ido A, Sato T, Nakashima D, Ueshima K, Ikeda M, Okusaka T, Tamura K, Furuse J. A randomized, double-blind, placebo-controlled, phase 3 study of tivantinib in Japanese patients with MET-high hepatocellular carcinoma. Cancer Sci. 2020 Oct;111(10):3759-3769. doi: 10.1111/cas.14582. Epub 2020 Aug 26. PMID 32716114